CLINICAL TRIAL: NCT05345743
Title: The Incidence of Postoperative Pulmonary Complications in Patients With a Positive and Negative AIR-Test During General Anesthesia
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr., Amsterdam UMC, location AMC
Other Study IDs: W22_079
Record Dates: First submitted 2022-04-11; First posted 2022-04-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Surgery--Complications; Atelectasis; Anesthesia
Keywords: Anesthesia; AIR-test; Postoperative Pulmonary Complications
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive AIR-test: Patients with a positive intraoperative AIR-test result
  Interventions: Procedure: Surgery
- Negative AIR-test: Patients with a negative intraoperative AIR-test result
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — All types of surgery requiring general anesthesia

SUMMARY:
The overall objective of this study is to describe the incidence of postoperative pulmonary complications in patients with a positive and negative AIR-test result. Second, the investigators wish to describe the incidence of a positive AIR-test and its association with the development of PPC. In addition, the investigators aim to describe whether mechanical ventilation strategy differs between patients with a positive and negative AIR-test.

DETAILED DESCRIPTION:
The 'AIR-test', a method wherein inspiratory oxygen concentration is reduced to 21% and pulse-oximetry hemoglobin saturation (SpO2) is monitored, can be used to demonstrate the presence of an atelectasis-induced alveolar shunt. It remains uncertain whether an intraoperative positive AIR-test is associated with clinical outcomes. It is hypothesized that in a general surgical population, the incidence of postoperative pulmonary complications (PPC) is higher in patients with a positive AIR-test than in patients with a negative AIR-test. The aim of this study is to describe the incidence of PPC in patients with a positive and in patients with a negative AIR-test. Second, the investigators want to describe the incidence of a positive AIR-test and its association with the development of PPC. The investigators also want to evaluate whether mechanical ventilation strategy differs between patients with a positive and negative AIR-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery under general anesthesia in the Amsterdam University Medical Centers, location Meibergdreef with an Endotracheal Tube;
* Patients > 18 years;
* Preoperative SpO2 of ≥97%;
* AIR-test performed after induction of anesthesia, in a hemodynamic and respiratory steady state.

Exclusion Criteria:

* Age < 18 years;
* No consent/objection;
* Patient participated in another conflicting interventional study on mechanical ventilation during general anesthesia

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgery under general anesthesia in whom an AIR test is performed
Sampling Method: Probability Sample
Enrollment: 632 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative pulmonary complications | The first 5 postoperative days
  Respiratory failure; Bronchospasm; Acute Respiratory Distress Syndrome (ARDS); Suspected pulmonary infection; Aspiration pneumonitis; Atelectasis; Pleural effusion; Pulmonary infiltrate; Cardiopulmonary effusion; Pneumothorax

SECONDARY OUTCOMES:
AIR-test result | Intraoperative period
  Number of patients with a positive and negative AIR-test
Tidal volume during general anesthesia for surgery | Intraoperative period
  Tidal volume in mL per kg predicted bodyweight
Positive End-Expiratory Pressure during general anesthesia for surgery | Intraoperative period
  Positive End-Expiratory Pressure in Centimeters of Water (cmH2O)
Peak Pressure during general anesthesia for surgery | Intraoperative period
  Peak Pressure in cmH20
Driving Pressure during general anesthesia for surgery | Intraoperative period
  Driving Pressure in cmH2O
Fraction of Inspired Oxygen during general anesthesia for surgery | Intraoperative period
  Fraction of Inspired Oxygen
End-tidal Carbon Dioxide (CO2) during general anesthesia for surgery | Intraoperative period
  End-tidal CO2 in millimeters of mercury (mmHg)
Respiratory Rate during general anesthesia for surgery | Intraoperative period
  Respiratory Rate per minute
The incidence of the individual components of postoperative pulmonary complications | The first 5 postoperative days
  Respiratory failure; Bronchospasm; ARDS; Suspected pulmonary infection; Aspiration pneumonitis; Atelectasis; Pleural effusion; Pulmonary infiltrate; Cardiopulmonary effusion; Pneumothorax
Length of hospital stay | From the day of surgery until the day of discharge, up to day 30
  Days of hospital stay
Rate of all-cause mortality and in-hospital mortality | Postoperative day 5 and postoperative day 30
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, Professor, Principal Investigator — Anesthesiology and Pain Medicine, AUMC location AMC; Marcus J Schultz, Professor, Principal Investigator — Intensive Care, AUMC location AMC
Locations (1):
- Amsterdam University Medical Centers, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hol L, Vermeulen TD, de Kruijk RS, Tjikhoeri A, Koning GRM, Breel JS, van Meenen DMP, Hollmann MW, Schultz MJ. Associations of a positive intra-operative air-test with postoperative pulmonary complications in general surgery patients: A single-centre prospective observational study. Eur J Anaesthesiol. 2025 Oct 23. doi: 10.1097/EJA.0000000000002304. Online ahead of print. PMID 41222052